CLINICAL TRIAL: NCT03905538
Title: Evaluation of [18F]FLT PET/CT as an Early Predictor of Outcome in Pediatric Solid Tumors
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Laura Klesse, Associate Professor of Pediatrics Hematology/Oncology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2019-0627
Record Dates: First submitted 2019-03-08; First posted 2019-04-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]FLT-PET/CT Arm (Experimental): The experimental [18F]FLT-PET/CT will be completed before initiation of chemotherapy and prior to the third cycle (or month) of chemotherapy. Laboratory analysis and correlative radiology, as directed per clinical care based on the primary diagnosis, are required within 30 days of the baseline [18F]FLT PET/CT. Follow-up will comprise 24 months of standard practice treatment and follow up.
  Interventions: Drug: [18F]FLT-PET/CT

INTERVENTIONS:
Drug: [18F]FLT-PET/CT — Dose of 0.07 mCi/Kg [18F]FLT to max of 5 mCi (± 20%) will be given intravenously.

SUMMARY:
The experimental [18F]FLT-PET/CT will be completed before initiation of chemotherapy at either diagnosis or initiation of salvage chemotherapy at relapse and prior to the third cycle (or month) of chemotherapy. Laboratory analysis and correlative radiology, as directed per clinical care based on the primary diagnosis, are required within 30 days of the baseline [18F]FLT PET/CT. Follow-up will comprise 24 months of standard practice treatment and follow up.

DETAILED DESCRIPTION:
Primary Objective is to assess if percentage change in [18F]FLT PET/CT quantitative parameters (SUV max, or SUV peak or proliferative tumor volume) after 2 cycles of chemotherapy can predict progression free survival at 1 and 2 years in pediatric patients with newly diagnosed or relapsed solid tumors.

Secondary Objectives are: (1) to assess if percentage change in [18F]FLT PET/CT quantitative parameters (SUV max, or SUV peak or proliferative tumor volume) after 2 cycles of chemotherapy can predict overall survival at 2 years in pediatric patients with newly diagnosed or relapsed solid tumors; and (2) for enrolled patients that undergo tumor resection as part of their therapy regimen within one month of the FLT imaging, mitotic index of the tumor will be assessed as compared to initial biopsy specimen and correlate with FLT activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed solid tumor malignancies with residual tumors present that require standard of care chemotherapy for a minimum number of cycles. All anatomical sites and all tumor histologies are eligible including central nervous system tumors. Both newly diagnosed and/or newly relapsed patients are eligible.
* Patients ages 8 - 25 years
* In the opinion of the investigator, patients must be thought to be able to lie still for imaging without sedation for 20 - 30 minutes.
* Patients must have a performance status of > 50% (Lansky or Karnofsky).
* Patients of childbearing potential must have a negative urine or serum pregnancy test as per institution's standard of care within 7 days prior to [18F]FLT PET/CT imaging.
* Ability to understand and the willingness to sign a written informed consent/assent.

Exclusion Criteria:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals of similar chemical or biologic composition to [18F]FLT
* Newly diagnosed subjects who had prior chemotherapy or radiotherapy before enrollment in the study. Relapsed patients are eligible prior to starting their relapsed chemotherapy regimen if they meet the other eligibility criteria.
* Subjects for whom chemotherapy is not a standard of care primary therapy option.
* Patients who are pregnant or breast-feeding.
* Patients with no residual tumor (i.e. complete resection at diagnosis or relapse).

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between change in [18F]FLT PET/CT and progression free and overall survival | up to 24 months following treatment
  Determine that a positive response (decrease in quantitative parameters) at an interim [18F]FLT PET/CT is related to progression free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Laura Klesse, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States